CLINICAL TRIAL: NCT00266305
Title: Fish Oil Supplementation in Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Research Agency (Other); BASF (Industry); Technical University of Denmark (Other)
Responsible Party: Associate profesor lotte lauritzen, Dept. of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KVL-IHE-D72; FØTEK 2: 93s-2468-å96-00020; FØTEK 3: 2011-00-0028; KF 01-300/98; KF 01-183/01
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Development and Health
Keywords: n-3 LCPUFA; Infant development; Visual acuity; Immune function; Breast milk
MeSH Terms: interventions — Fish Oils

ARMS (3):
- Fish oil (Experimental)
  Interventions: Behavioral: Fish oil (Dry n-3, BASF)
- Olive oil (Placebo Comparator): Control group
  Interventions: Behavioral: Fish oil (Dry n-3, BASF)
- High fish (No Intervention): Reference group

INTERVENTIONS:
Behavioral: Fish oil (Dry n-3, BASF) — 5 g/oil daily for the first four month of lactation
  Arms: Fish oil; Olive oil

SUMMARY:
The main purpose of the study was to examine whether fish oil supplementation of lactating mothers affect infant development during first year of life, focusing on visual and mental development. A follow-up studies are conducted in order to see if early intake of long-chain n-3 polyunsaturated fatty acids (n-3 LCPUFA) have any long-term effects on health, primarily immun function and markers of cardiovascular risk.

DETAILED DESCRIPTION:
Background:

Studies indicate that infants, who are fed formula without n-3 LCPUFA, have slower visual development than those, who receive n-3 LCPUFA in breast-milk. The mental development seems also to depend on whether infants are breast-fed or not. Long-term health has also been proposed to be affected (The infant origin of adult disease hypothesis). It is not clear whether these differences is due to dietary LCPUFA as comparison of breast-fed and formula-fed infants are complicated by the socio-demographic differences that exist between mother, who choose to breast-feed or not. Recent studies indicate that LCPUFA supplementation of formulas has beneficial effects on the visual acuity and mental abilities of infants. The LCPUFA content of breast-milk varies and this could potentially be of importance for infant development.

Methods:

211 pregnant women with a high (>80 percentile) or low (< mean) fish intake were recruited. After birth mother with low fish intake were randomized to receive 4 g/day of fish oil or olive oil for the first 4 months of the lactation period. 150 mother-infant pairs were followed for 1 year gathering information on maternal n-3 LCPUFA intake and infant development (growth, developmental milestones, visual acuity, cognitive functions and language acquisition). Milk samples were collected at 0, 2, 4 and 9 months and blood samples were taken from the mother and the infant at 4 months of age in order to determine the biochemical effect of the supplementation.

The children were followed-up at 2½ years of age and around 7 years of age. The study is performed in association to the National Birth Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with uncomplicated singleton pregnancy
* No metabolic disorders and prepregnancy BMI < 30 kg/m2
* Intention to exclusively breast-feed for 4 mo
* Fish intake below the Danish mean or above 80th percentile (reference group)

Exclusion Criteria:

* Pre- or post term delivery (< 37 or > 43 wks of gestation)
* Abnormal weight for gestation (outside 10th-90th percentile range)
* Apgar score 5 min after delivery < 8
* Infant admission to a neonatal department
* If supplementation did not begin within 2 wks after delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1998-12; Study Completion 2007-01

PRIMARY OUTCOMES:
Breast milk fatty acid composition - 0, 2, 4 and 9 mo
Fatty acid composition of infant RBC at 4 mo
Visual acuity - 2 and 4 mo
Follow-up:
Anthropometric measures
Blood pressure
Ex vivo cytokine production (e.g. IL-10 and interferon-γ) in whole blood after 24 h of stimulation with bacterial components

SECONDARY OUTCOMES:
Anthropometric measures - 0, 2, 4 and 9 mo
Problem solving at 9 mo
Language development (CDI) at 1 and 2 y
Contrast sensitivity at 2 mo
Vernier acuity at 4 mo
Follow-up:
Heart rate variability
Endothelial function measured by PWV
Plasma IgE
Diet
RBC fatty acid composition
Plasma growth factors

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, Ph.D, Principal Investigator — Department of Human Nutrition, Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Result] Lauritzen L, Jorgensen MH, Mikkelsen TB, Skovgaard lM, Straarup EM, Olsen SF, Hoy CE, Michaelsen KF. Maternal fish oil supplementation in lactation: effect on visual acuity and n-3 fatty acid content of infant erythrocytes. Lipids. 2004 Mar;39(3):195-206. doi: 10.1007/s11745-004-1220-8. PMID 15233397
- [Result] Lauritzen L, Hoppe C, Straarup EM, Michaelsen KF. Maternal fish oil supplementation in lactation and growth during the first 2.5 years of life. Pediatr Res. 2005 Aug;58(2):235-42. doi: 10.1203/01.PDR.0000169978.92437.58. Epub 2005 Jul 8. PMID 16006428
- [Result] Hoppe C, Udam TR, Lauritzen L, Molgaard C, Juul A, Michaelsen KF. Animal protein intake, serum insulin-like growth factor I, and growth in healthy 2.5-y-old Danish children. Am J Clin Nutr. 2004 Aug;80(2):447-52. doi: 10.1093/ajcn/80.2.447. PMID 15277169
- [Result] Ulbak J, Lauritzen L, Hansen HS, Michaelsen KF. Diet and blood pressure in 2.5-y-old Danish children. Am J Clin Nutr. 2004 Jun;79(6):1095-102. doi: 10.1093/ajcn/79.6.1095. PMID 15159241
- [Result] Lauritzen L, Kjaer TM, Fruekilde MB, Michaelsen KF, Frokiaer H. Fish oil supplementation of lactating mothers affects cytokine production in 2 1/2-year-old children. Lipids. 2005 Jul;40(7):669-76. doi: 10.1007/s11745-005-1429-6. PMID 16196417
- [Result] Lauritzen L, Jorgensen MH, Olsen SF, Straarup EM, Michaelsen KF. Maternal fish oil supplementation in lactation: effect on developmental outcome in breast-fed infants. Reprod Nutr Dev. 2005 Sep-Oct;45(5):535-47. doi: 10.1051/rnd:2005044. PMID 16188206
- [Result] Larnkjaer A, Christensen JH, Michaelsen KF, Lauritzen L. Maternal fish oil supplementation during lactation does not affect blood pressure, pulse wave velocity, or heart rate variability in 2.5-y-old children. J Nutr. 2006 Jun;136(6):1539-44. doi: 10.1093/jn/136.6.1539. PMID 16702318